CLINICAL TRIAL: NCT00502294
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled, Multicenter Study of Visilizumab in Subjects With Intravenous Steroid-Refractory Ulcerative Colitis
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Facet Biotech (Industry)
Collaborators: PDL BioPharma, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 291-416
Record Dates: First submitted 2007-07-13; First posted 2007-07-17 (Estimated); Last update posted 2009-06-25 (Estimated); Status verified 2008-07

CONDITIONS: Intravenous Steroid-Refractory Ulcerative Colitis
Keywords: Ulcerative Colitis, UC, Intravenous Steroid-Refractory Ulcerative Colitis, IVSR-UC
MeSH Terms: conditions — Colitis, Ulcerative | interventions — visilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Visilizumab (HuM291; Nuvion®)

SUMMARY:
To compare the efficacy of visilizumab at 5 mcg/kg/day administered intravenously (IV) on Days 1 and 2 to placebo in subjects with IVSR-UC.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, 18 years of age or older.
* Diagnosis of UC verified by endoscopy within 60 months prior to consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)